CLINICAL TRIAL: NCT05862402
Title: Dose Optimization by PK/PD of Antibiotics to Improve Clinical Outcome of CRKP Bloodstream Infections in Critically Ill Patients and in Vitro Study of Monotherapy, Combination Therapy and Molecular Biology of Drug Resistance at Phramongkutklao Hospital: Prospective, Historical Controlled Study
Brief Title: Dose Optimization by Pharmacokinetic/Pharmacodynamic of Antibiotics to Improve Clinical Outcome of Carbapenem Resistant Klebsiella Pneumoniae Bloodstream Infections in Critically Ill Patients at Phramongkutklao Hospital
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Collaborators: Silpakorn University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMK-0008
Record Dates: First submitted 2023-04-26; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Carbapenem Resistant Klebsiella Pneumoniae
Keywords: Antibiotics; Dose optimization; Clinical outcome; CRKP; Critically ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Prospective study compare historical controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Dose antibiotics adjusted by pharmacokinetic and pharmacodynamic using Monte Carlo simulation
  Interventions: Drug: Dose-adjustment by PKPD
- Control group (No Intervention): Dose antibiotics from standard care

INTERVENTIONS:
Drug: Dose-adjustment by PKPD — Dose-adjustment by pharmacokinetic and pharmacodynamic using Monte Carlo simulation
  Other Names: Antibiotics: Ceftazidime-Avibactam or Combination antibiotics (eg. Meropenem-Colistin, Imipenem-Colistin, Tigecycline-Amikacin, Tigecycline-Gentamicin, Tigecycline-Meropenem or Tigecycline-Colistin)
  Arms: Intervention group

SUMMARY:
The patients who infected with Carbapenem resistant Klebsiella pneumoniae were high mortality rate. Appropriate antibiotics therapy adjusted by Pharmacokinetic/Pharmacodynamic plays an important role in determining outcomes in Critically ill patients. Consequently, standard antibiotics dose may not be adequate to achieve pharmacokinetic/pharmacodynamic target in Critically ill patients. The purpose of this study is to compare the clinical outcomes between the critically ill patients who received antibiotics dose adjusted by pharmacokinetic/pharmacodynamic using Monte Carlo simulation and historical critically ill patients who received antibiotics from standard practice.

ELIGIBILITY:
Inclusion Criteria:

1. 20 years and older who admitted at Phramongkutklao Hospital
2. Patients who was diagnosed blood stream infection with CRKP between April 10th, 2023 to March 31st, 2024 (Prospective study) and January 1st, 2012 to March 31st, 2023 (Retrospective study); Historical group
3. Patients who had signs and symptoms at least 1 criteria following:

   3.1. Patients who had signs and symptoms of Systemic Inflammatory Response Syndrome (SIRS) at least 2 criteria:
   * Temperature above 38 oC or below 36 oC
   * Heart rate more than 90 beats/min
   * Respiratory rate more than 20 /min or PaCO2 less than 32 mmHg (4.3 kPa)
   * White blood cell more than 12,000 cell/mm3 or less than 4,000 cell/mm3 3.2. Patients who was diagnosed sepsis or SOFA score or qSOFA score at least 2 score 3.3. Patients who was diagnosed septic shock or who had hypotension with adequate fluid and need for vasopressor to maintain mean arterial pressure over 65 mmHg and serum lactate above 2 mmol/L
4. Patients who received antibiotics at least 48 hours which are as follow:

   * Ceftazidime-Avibactam or
   * Combination antibiotics (eg. Meropenem-Colistin, Imipenem-Colistin, Tigecycline-Amikacin, Tigecycline- Gentamicin, Tigecycline-Meropenem or Tigecycline-Colistin)

Exclusion Criteria:

1. Patients who were pregnancy or breastfeeding
2. Patients who had drug allergy (eg. Ceftazidime-Avibactam, Tigecycline, Amikacin, Gentamicin, Imipenem, Meropenem or Colistin)
3. Patients who not to received resuscitation.
4. Patients who were end stage cancer.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-05-07 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | 14 day
  Alive or death

SECONDARY OUTCOMES:
Mortality | 30 days
  Alive or death
Microbiological cure rate | 14 days
  Evaluated culture of bloodstream
Hospital length of stay | With in 30 days
  Time interval (day) from hospital admission (after enrolled) to hospital discharge or death from any cause
ICU length of stay | With in 30 days
  Time interval (day) from ICU admission (after enrolled) to ICU discharge or death from any cause
Clinical cure rate | Through treatment completion or with in 30 days
  Evaluated sign and symptoms of infection or culture no growth
Duration of vasopressor or Inotropic agents | With in 30 days
  Time interval (day) from time of vasopressor or Inotropic agents initiation to time to vasopressor or Inotropic agents discontinuation
Duration of ventilator | Assessed with in 30 days
  Time interval (day) of ventilator
Ventilator free day | 30 days
  Day alive and free of ventilator
Vasopressor or Inotropic drug free day | 30 days
  Day alive and free of vasopressor or inotropic drug
Procalcitonin | 14 days
  Evaluated serum procalcitonin
Adverse event | Day 0, 5, 7 and finish course of Antibiotics or discharge
  Evaluated side effect (eg. seizure, liver impairment, renal impairment)

CONTACTS AND LOCATIONS:
Overall Officials: Sujareenoot Suya, PharmD, Study Chair — Faculty of Pharmacy, Silpakorn University; Weerayuth Saelim, BCP, Study Director — Faculty of Pharmacy, Silpakorn University; Wichai Santimaleeworagun, PhD, Study Director — Faculty of Pharmacy, Silpakorn University; Worapong Nasomsong, MD, Study Director — Phramongkutklao College of Medicine and Hospital
Locations (1):
- Phramongkutklao Hospital, Ratchathewi, Bangkok, Thailand